CLINICAL TRIAL: NCT03503500
Title: Effectiveness of a Laid-back Breastfeeding Approach on Breastfeeding Initiation in Hospital Setting. A Randomized Controlled Trial
Brief Title: Laid-back Breastfeeding in Hospital Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC 29/17
Record Dates: First submitted 2018-03-28; First posted 2018-04-19 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Laid-back position; Breast problems; Exclusive breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Open label, randomized parallel controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laid-back breastfeeding (Experimental): Women will breastfed in relaxed, laid-back position, with her baby laying prone on her, so that the baby's body is in the largest possible contact with mother's curves, without following particular procedure to breastfed.
  Interventions: Other: Laid-back breastfeeding
- Standard care (Active Comparator): Staff will show to mothers how to breastfeed and will help them to attach the baby correctly to the breast,
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Laid-back breastfeeding — At randomization the Italian version of the video "Biological nurturing", which provides detailed information on LB BF, will be delivered to women with the recommendation to watch it before birth; during the maternity ward stay, adequately trained staff will support women to breastfed in relaxed, laid-back position, with her baby laying prone on her, so that the baby's body is in the largest possible contact with mother's curves. In the maternity ward a daily supervision by an external expert on LB BF will be provided
  Arms: Laid-back breastfeeding
Other: Standard care — 2. the standard care in use at the Institute (WHO/UNICEF 20-hours course) (control group). At randomization, the Italian version of the video "Breast is best" (Allattare informati), which provides detailed information on standard support to breastfeeding, will be delivered to women with the recommendation to watch it before birth; during the maternity ward stay, the staff will show to mothers how to breastfeed and will help them to attach the baby correctly to the breast
  Arms: Standard care

SUMMARY:
The so-called biological nurturing (BN) - or laid-back breastfeeding (LB BF), a new neurobehavioral approach to breastfeeding (BF), has the potential to enhance BF initiation and to reduce breast problems (pain, fissures, etc.), while easing the newborn attachment to the breast. BN focuses on facilitating the mother to breastfeed in a relaxed, laid-back position, with her baby laying prone on her, so that the baby's body is in the largest possible contact with mother's curves. This position opens up the mother's body and promotes baby's movements through the activation of 20 primary neonatal reflexes stimulating BF. Neurophysiological studies show that, through this approach, infants instinctively know how to feed, thanks to the presence of neonatal reflexes, at the same time mothers being able to instinctively activate the same reflexes.

The main objective of this study is to assess the effectiveness of LB BF compared to standard hospital practices on the frequency of breast problems (i.e., pain, fissures, etc.) at discharge.

DETAILED DESCRIPTION:
Despite the fact that breastfeeding (BF) benefits are largely known and that this practice is highly recommended, available data at national and international level show that exclusive breastfeeding rates are still low. Among the main determinants that can be addressed to improve BF prevalence, the quality of care and the support provided by health staff to women during labour and delivery seem to have a particular relevance. In hospital settings, an adequate support to women initiating BF is not always granted, especially where time availability of staff is limited and their specific skills inadequate.

In most recent years, a growing scientific evidence on neonatal primary reflexes opened new windows of intervention. In particular, the so-called biological nurturing (BN) - or laid-back breastfeeding (LB BF) - has the potential to enhance BF initiation and to reduce breast problems (pain, fissures, etc.), while easing the newborn attachment to the breast. BN is a new neurobehavioral approach to BF initiation, which focuses on facilitating the mother to breastfeed in a relaxed, laid-back position, with her baby laying prone on her, so that the baby's body is in the largest possible contact with mother's curves. This position opens up the mother's body and promotes baby's movements through the activation of 20 primary neonatal reflexes stimulating BF. Neurophysiological studies show that, through this approach, infants instinctively know how to feed, thanks to the presence of neonatal reflexes, at the same time mothers being able to instinctively activate the same reflexes.

The method is simple, given that there are no "correct" positions nor the need to follow particular procedures to BF, whilst with the traditional approach precise indications on the right BF position and attachment are to be provided to and followed by the woman. The effectiveness of BN has however not been adequately studied through randomized controlled trials, particularly in hospital settings.

The main objective of this study is to assess the effectiveness of LB BF compared to standard hospital practices on the frequency of breast problems (i.e., pain, fissures, etc.) at discharge. Secondary study objectives are to assess the effectiveness of the intervention on: exclusive breastfeeding at discharge and during the maternity ward stay; exclusive breastfeeding at 7 days and 1 and 4 months of life; frequency of breast problems at 7 days and 1 and 4 months of life; frequency of use of nipple shield at discharge, at 7 days, and at 1 and 4 months. Furthermore, the study will assess the feasibility of the LB BF approach in hospital setting and the degree of mother satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* women who plan to give birth at the Institute for Maternal and Child Health Burlo Garofolo, Trieste, and who express the intention to breastfeed, identified during the visit for their 3rd routine antenatal ultrasound scan (30/32 weeks gestational age).

Exclusion Criteria:

* presence of problems with potential negative impact on BF (e.g. severe cardiovascular problems, severe obesity as defined by body mass index above 32; hypertensive disorders);
* antenatal diagnosis of foetal complex diseases (i.e., congenital pulmonary adenomatoid malformation);
* twin pregnancy. The need for admission at birth or during hospital stay to Intensive Care Unit of both newborn or mother and the appearance of pathological jaundice in newborn are reasons for exclusion after randomization.

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 208 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Breast problems | Within 7 days of birth, at discharge from hospital
  Frequency of breast problems (i.e., pain, fissures, etc.) during the hospital stay

SECONDARY OUTCOMES:
Breast problems | 7 days after discharge from hospital
  Frequency of breast problems (i.e., pain, fissures, etc.)
Breast problems | 30 days after discharge from hospital
  Frequency of breast problems (i.e., pain, fissures, etc.)
Breast problems | 120 days after discharge from hospital
  Frequency of breast problems (i.e., pain, fissures, etc.)
Exclusive breastfeeding during the hospital stay | Within 7 days of birth, at discharge from hospital
  Frequency of exclusive breastfeeding (according to the World Health Organization definitions) during the hospital stay
Exclusive breastfeeding in the last 24 hours of hospital stay | Within 7 days of birth, at discharge from hospital
  Frequency of exclusive breastfeeding (according to the World Health Organization definitions) in the last 24 hours of hospital stay
Exclusive breastfeeding | 7 days after discharge from hospital
  Frequency of exclusive breastfeeding (according to the World Health Organization definitions)
Exclusive breastfeeding | 30 days after discharge from hospital
  Frequency of exclusive breastfeeding (according to the World Health Organization definitions)
Exclusive breastfeeding | 120 days after discharge from hospital
  Frequency of exclusive breastfeeding (according to the World Health Organization definitions)
Use of nipple shield | Within 7 days of birth, at discharge from hospital
  Frequency of use of nipple shield
Use of nipple shield | 7 days after discharge from hospital
  Frequency of use of nipple shield
Use of nipple shield | 30 days after discharge from hospital
  Frequency of use of nipple shield
Use of nipple shield | 120 days after discharge from hospital
  Frequency of use of nipple shield
Mother satisfaction | Within 7 days of birth, at discharge from hospital
  Degree of maternal satisfaction evaluated using the specific subscale of the Maternal Breastfeeding Evaluation Scale (MBFES). MBFES is a 30 item scale that measures the mother's evaluation of breastfeeding, with answers given on a 5 point Likert scale (1=strongly disagree to 5=strongly agree). For the purpose of this study, only the Maternal Enjoyment/Role Attainment Subscale (questions 1, 2, 6, 9, 11, 12, 16, 17, 18, 20, 21, 23, 25, and 30) will be used
Mother satisfaction | 30 days after discharge from hospital
  Degree of maternal satisfaction evaluated using the specific subscale of the Maternal Breastfeeding Evaluation Scale (MBFES). MBFES is a 30 item scale that measures the mother's evaluation of breastfeeding, with answers given on a 5 point Likert scale (1=strongly disagree to 5=strongly agree). For the purpose of this study, only the Maternal Enjoyment/Role Attainment Subscale (questions 1, 2, 6, 9, 11, 12, 16, 17, 18, 20, 21, 23, 25, and 30) will be used
Mother satisfaction | 120 days after discharge from hospital
  Degree of maternal satisfaction evaluated using the specific subscale of the Maternal Breastfeeding Evaluation Scale (MBFES). MBFES is a 30 item scale that measures the mother's evaluation of breastfeeding, with answers given on a 5 point Likert scale (1=strongly disagree to 5=strongly agree). For the purpose of this study, only the Maternal Enjoyment/Role Attainment Subscale (questions 1, 2, 6, 9, 11, 12, 16, 17, 18, 20, 21, 23, 25, and 30) will be used
Feasibility of the LB BF approach in hospital setting | Within 7 days of birth, at discharge from hospital
  Frequency of women who do not consent to participate or who withdraw from the study or who crossover between groups or who receive a different intervention from that allocated

CONTACTS AND LOCATIONS:
Overall Officials: Luca Ronfani, MD, Study Director — IRCCS Burlo Garofolo, Trieste, Italy; Mariarosa Milinco, BF counselor, Principal Investigator — IRCCS Burlo Garofolo, Trieste, Italy
Locations (1):
- Institute for Maternal and Child Health IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Milinco M, Travan L, Cattaneo A, Knowles A, Sola MV, Causin E, Cortivo C, Degrassi M, Di Tommaso F, Verardi G, Dipietro L, Piazza M, Scolz S, Rossetto M, Ronfani L; Trieste BN (Biological Nurturing) Investigators. Effectiveness of biological nurturing on early breastfeeding problems: a randomized controlled trial. Int Breastfeed J. 2020 Apr 5;15(1):21. doi: 10.1186/s13006-020-00261-4. PMID 32248838